CLINICAL TRIAL: NCT03753737
Title: A Study of the Relationship Between Personality Disorders and Substance Use Disorders in a Sexual Context in the Man Having Sex With Other Men Population - An Observational Study Based on a Cross-sectional Survey.
Brief Title: Personality Disorders and Substance Use Disorders in a Sexual Context in the Man Having Sex With Other Men Population
Acronym: PSYCHEMS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0509; 2018-A02168-47 (Other: ID-RCB)
Record Dates: First submitted 2018-11-22; First posted 2018-11-27 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemsex: Men who have Sex with Men (MSM) attending an addiction care center for past or present mild, moderate or severe substance-related disorder(s) according to DSM-V criteria, occurring in a sexual context and concerning cathinones, GHB/GBL, methamphetamine, cocaine and/or ketamine.
  Interventions: Other: Questionnaires and semi-structured interview
- Control: Men who have Sex with Men (MSM) consulting for a PrEP (HIV Pre-Exposure Prophylaxis) prescription who have never used cathinones, GHB/GBL, methamphetamine, cocaine or ketamine before or during sex.
  Interventions: Other: Questionnaires and semi-structured interview

INTERVENTIONS:
Other: Questionnaires and semi-structured interview — * Questionnaires : PDQ-4+ (personality disorders), HAD (Anxiety and Depression), AUDIT-c (Alcohol consumption), CTQ-SF (Childhood Trauma Questionnaire).
  * Semi-structured interview : Evaluation of socio-demographic characteristics, psychiatric and addiction comorbidities, sexually transmitted infections, sexual practices, sexual dysfunction, hypersexual disorder.

SUMMARY:
Chemsex refers to the use of psychoactive drugs in a sexual context, mainly cathinones, GHB/GBL, methamphetamine, cocaine and ketamine. This can cause infectious or psychiatric complications, addictions, and often goes with high risk sexual behaviours. Recent studies have highlighted the relationship between personality disorders, substance use disorders and risky sexual behaviours. It is important to understand the factors associated with chemsex in order to offer adapted prevention and care plans.

The study hypothesis is that personality disorders, evaluated with the PDQ-4+ questionnaire, are more frequent among man having sex with other men with a substance use disorder linked to chemsex than among man having sex with other men who have never practised chemsex.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Men who have Sex with Men
* No opposition to participate to the study
* Chemsex group: to attend an addiction care center for past or present mild, moderate or severe substance-related disorder(s) according to DSM-V criteria, occurring in a sexual context and concerning cathinones, GHB/GBL, methamphetamine, cocaine and/or ketamine.
* Control group: to consult for a PrEP prescription and never have used cathinones, GHB/GBL, methamphetamine, cocaine or ketamine before or during sex.

Exclusion Criteria:

* Deprivation of liberty
* Guardianship
* Chemsex group: simple experience of chemsex without substance use disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Men who have Sex with Men (MSM) with past or present substance-related disorder related to chemsex, and sexually active MSM who have never experienced chemsex.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Personality disorders | 1 day
  Positive score for 1 or more DSM-V personality disorders(PD) using French version of the PDQ4+,Personality Diagnostic Questionnaire-Version4,comprising:
  * Combined score of overall personality disturbance (ranges0 to 93);higher values reflect a more important personality disturbance
  * Borderline PD:Score Ranges(SR) 0 to 9,positive(+) if ≥ 5
  * Narcissistic PD:SR 0 to 9,+ if ≥5
  * Histrionic PD:SR 0 to 8,+ if ≥5
  * Antisocial PD:SR 0 to 8,+ if ≥4 and criteria 99 positive
  * Avoidant PD:SR 0 to 7,+ if ≥4
  * Dependent PD:SR 0 to 8,+ if ≥5
  * Obsessive-Compulsive PD:SR 0 to 8,+ if ≥4
  * Paranoid PD:SR 0 to 7,+ if ≥4
  * Schizoid PD:SR 0 to 7,+ if ≥4
  * Schizotypal PD:SR 0 to 9,+ if ≥5
  * Questionnaire must be interpreted with caution if 1 of the 2 "Suspect Questionnaire" items is +, or if at least 2 of the 4 "Too Good" items are +
  * Negativistic and depressive PD are evaluated with the PDQ4+ but are not part of the outcome measures in the study

CONTACTS AND LOCATIONS:
Locations (1):
- CSAPA - Service Hépato-gastroentérologie, Lyon, France

IPD SHARING:
Plan to Share IPD: No